CLINICAL TRIAL: NCT04348851
Title: Internet and Telephone Support Intervention for Stroke Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1395-P
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Depression; Quality of Life; Recovery of Function; Self Efficacy; Stress
Keywords: stroke; caregiving
MeSH Terms: conditions — Depression; Stroke

STUDY DESIGN:
Intervention Model Description: Four-arm randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigator and staff collecting outcome data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 4-Week Intervention (Experimental): Registered nurses (RNs) will conduct the combined Internet and telephone intervention condition. The intervention is based on the relational/problem-solving model of stress originally developed by D-Zurilla and Nezu. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on our national RESCUE Stroke Caregiver website. (http://www.cidrr8.research.va.gov/rescue/).
  Interventions: Behavioral: Caregiver problem-solving
- 8-Week Intervention (Experimental): Registered nurses (RNs) will conduct the combined Internet and telephone intervention condition. The intervention is based on the relational/problem-solving model of stress originally developed by D-Zurilla and Nezu. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on our national RESCUE Stroke Caregiver website. (http://www.cidrr8.research.va.gov/rescue/).
  Interventions: Behavioral: Caregiver problem-solving
- 8-Week Attention Control (Active Comparator): The Registered Nurses (RNs) will only provide active listening and paraphrasing. The RNs will ask caregivers to talk about their caregiver experiences. The nurses will not provide advice, but rather direct caregivers to access information on the Caregiver Family Alliance website (www.caregiver.org) for managing problems or to contact their healthcare provider.
  Interventions: Behavioral: Attention Control
- Standard Care (No Intervention): Caregivers receiving standard of care

INTERVENTIONS:
Behavioral: Caregiver problem-solving — Registered nurses will conduct the combined Internet and telephone intervention condition. The intervention is based on the relational/problem-solving model of stress originally developed by D-Zurilla and Nezu. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on our national RESCUE Stroke Caregiver website. (http://www.cidrr8.research.va.gov/rescue
  Arms: 4-Week Intervention; 8-Week Intervention
Behavioral: Attention Control — The RNs will only provide active listening and paraphrasing. The RNs will ask caregivers to talk about their caregiver experiences. The nurses will not provide advice, but rather direct caregivers to access information on the Caregiver Family Alliance website (www.caregiver.org) for managing problems or to contact their healthcare
  Arms: 8-Week Attention Control

SUMMARY:
This study will test a problem-solving and support intervention for caregivers of veterans with stroke. The investigators will assign caregivers to one for four groups: 4-session intervention, 8-session intervention, attention control (active listening), or standard care. The investigators will assess the impact of the intervention on caregiver outcomes (depression, burden, stress, problem-solving abilities, self-efficacy, and quality of life) and veteran outcomes (functional abilities).

DETAILED DESCRIPTION:
Background: Caregiver depression and burden are common following a family member's stroke and are major contributors of stroke survivors' functional recovery, resource use, and institutionalization. Previous studies reveal that problem-solving interventions are effective in improving caregiver and Veteran outcomes post-stroke. However, most of these studies were burdensome for caregivers and labor intensive because they involved multiple, face-to-face sessions. To overcome this shortcoming, the long-term goal is to implement caregiver programs that involve low-cost, evidence-based interventions that can be sustained in routine clinical practice. The investigators' immediate objective is to pilot test a problem-solving intervention that uses telephone support plus the Internet (i.e., the team's previously developed and nationally available RESCUE website) to improve the quality caregiving and the rehabilitation of Veterans. This pilot randomized controlled trial (RCT) simulates all aspects of a planned, future merit review proposal. This work builds on the team's extensive experience in caregiver education.

Aim #1: To explore the impact of a 4-session and 8-session Internet and telephone support intervention on stroke caregiver and Veteran outcomes when compared to an attention-control condition and standard care. The investigators will obtain preliminary data on effect estimates, group differences, and information on variability, correlations, and data ranges. Data will inform a sample size calculation for the larger trial and provide preliminary information on the impact of different doses of the intervention.

Aim #2: Determine caregivers' perceptions of the interventions and the attention control condition: Acceptability, facilitators/barriers, credibility of the nurse interventionists. The investigators will learn the strengths and weaknesses of the project, thereby helping to make improvements in the investigators' future merit project.

Methods: The investigators will conduct a four-arm, randomized controlled trial with three assessment points (baseline and two post-tests) and use mixed methods to determine caregivers' perceptions of the intervention and the attention control condition. The investigators will enroll 48 stroke caregivers whose Veterans receive care in VISN8. Eligible caregivers will complete baseline measures and then will be randomized to four arms: 1) 4-session intervention, 2) 8-session intervention, 3) attention control condition, or 4) standard care. Registered nurses will conduct the combined Internet and telephone intervention and the attention-control condition. The intervention is based on the relational/problem-solving model of stress originally developed by D-Zurilla and Nezu. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on the national RESCUE Stroke Caregiver website. (http://www.cidrr8.research.va.gov/rescue/). For the first post-test, a research team member will telephone caregivers to answer questions on instruments with established reliability and validity. A second post-test will be conducted approximately four to five months after the first post-test assessment to evaluate longer-term effects. Qualitative interviews will be conducted with 18 caregivers to obtain in-depth perceptions of the credibility of nurses, and value, facilitators, and barriers of the intervention and the attention control condition.

ELIGIBILITY:
Inclusion Criteria:

All non-paid caregivers of Veterans with a primary diagnosis of stroke, discharged to home from a medical or rehabilitation facility are eligible for participation if they meet the following criteria:

* have caregiving responsibility for a Veteran who has a diagnosis of stroke (ICD9 codes for stroke: 430-438) within the last 2.5 years and who have at least one activity of daily living (ADL), cognitive, or speech deficit related to stroke
* score 1 or greater on the Perceived Stress Scale
* have Internet access and ability
* are reachable by their cell or home phones
* read English at a seventh-grade reading level or better
* agree to random assignment to a study arm

Exclusion Criteria:

The investigators will exclude caregivers who fail to meet one or more of the inclusion criteria and whose Veterans:

* have a life expectancy of less than 6 months
* are receiving hospice/palliative care or are residing in a community living center

  * Life expectancy will be determined by reviewing the electronic health record (EHR) and conferring with our physician and clinical team members

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2016-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance R. Uphold, PhD MS BS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] LeLaurin J, Schmitzberger M, Eliazar-Macke N, Freytes IM, Dang S, Uphold C. A commentary on methodological issues in stroke caregiver research: lessons learned from three RESCUE intervention studies. Top Stroke Rehabil. 2019 Jul;26(5):399-404. doi: 10.1080/10749357.2019.1607485. Epub 2019 Apr 30. PMID 31038012

RESULTS

PARTICIPANT FLOW:
Groups:
- 4-Week Intervention; 8-Week Intervention: Registered nurses will conduct the combined Internet and telephone intervention condition. The intervention is based on the relational/problem-solving model of stress originally developed by D-Zurilla and Nezu. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on our national RESCUE Stroke Caregiver website. (http://www.cidrr8.research.va.gov/rescue/).
  Caregiver problem-solving: Registered nurses will conduct the combined Internet and telephone intervention condition. The intervention is based on the relational/problem-solving model of stress originally developed by D-Zurilla and Nezu. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on our national RESCUE Stroke Caregiver website. (http://www.cidrr8.research.va.gov/rescue
Period: Post-Test 1
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Started | 13 | 13 | 13 | 14
Completed | 13 | 11 | 13 | 14
Not Completed | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Post-Test 2
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Started | 13 | 11 | 13 | 14
Completed | 13 | 10 | 13 | 13
Not Completed | 0 | 1 | 0 | 1
Not completed — Stroke survivor death | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 8-Week Attention Control: The RNs will only provide active listening and paraphrasing. The RNs will ask caregivers to talk about their caregiver experiences. The nurses will not provide advice, but rather direct caregivers to access information on the Caregiver Family Alliance website (www.caregiver.org) for managing problems or to contact their healthcare provider.
  Attention Control: The RNs will only provide active listening and paraphrasing. The RNs will ask caregivers to talk about their caregiver experiences. The nurses will not provide advice, but rather direct caregivers to access information on the Caregiver Family Alliance website (www.caregiver.org) for managing problems or to contact their healthcare
- Total: Total of all reporting groups
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care | Total
Number analyzed (Participants) | 13 | 13 | 13 | 14 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.9) | 58.2 (12.0) | 57.1 (9.9) | 61.9 (9.5) | 60.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 12 | 12 | 49
  Male | 1 | 0 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 12 | 13 | 12 | 14 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 3 | 2 | 14
  White | 7 | 8 | 10 | 11 | 36
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 13 | 14 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms
Description: Changes in depressive symptoms will be measured with the Center for Epidemiologic Studies Depression (CES-D) scale. The CES-D is a 20-item, 4-point Likert scale ranging from never (0) to most of the time (3). Possible scores range from 0-60 with higher scores indicating more symptoms. It has been used in numerous studies with caregivers and has good reliability and validity.
Time Frame: 9 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 11 | 13 | 14
score on a scale | -2.31 (4.80) | 1.00 (7.52) | .08 (11.03) | 3.9 (8.66)

2. Primary Outcome: Change in Caregiver Burden
Description: Changes in burden will be measured by the Short Version of the Zarit Burden Interview (S-ZBI). This 12-item instrument was reduced from the original 29-item instrument. This instrument is scored on a 5-point Likert scale ranging from 0 (never) to 4 (nearly always). Possible scores range from 0-48 with higher scores indicating higher burden. The instrument was originally developed to measure dementia caregiver burden, but, the S-ZBI has been used in stroke caregiver studies and items are appropriate for other caregiver populations.
Time Frame: 9 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 11 | 13 | 14
score on a scale | -.92 (4.33) | .18 (3.34) | -.62 (7.03) | .14 (5.10)

3. Primary Outcome: Change in Depressive Symptoms
Description: Change in depressive symptoms will be measured with the Center for Epidemiologic Studies Depression (CES-D) scale. The CES-D is a 20-item, 4-point Likert scale ranging from never (0) to most of the time (3). Possible scores range from 0-60 with higher scores indicating more symptoms. It has been used in numerous studies with caregivers and has good reliability and validity.
Time Frame: 25 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 10 | 13 | 13
score on a scale | .92 (8.88) | -1.50 (4.58) | -3.46 (9.65) | 1.92 (4.87)

4. Primary Outcome: Change in Caregiver Burden
Description: Changes in burden will be measured by the Short Version of the Zarit Burden Interview. This 12-item instrument was reduced from the original 29-item instrument. This instrument is scored on a 5-point Likert scale ranging from 0 (never) to 4 (nearly always). Possible scores range from 0-48 with higher scores indicating higher burden. The instrument was originally developed to measure dementia caregiver burden, but, the S-ZBI has been used in stroke caregiver studies and items are appropriate for other caregiver populations.
Time Frame: 25 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 10 | 13 | 13
score on a scale | -.08 (5.36) | -.40 (5.52) | -.38 (5.39) | -.54 (3.5)

5. Secondary Outcome: Change in Health-Related Quality of Life - Physical Scale
Description: Changes in health-related quality of life will be measured by the Rand 12-item Health Survey (VR-12). The VR-12 items are scored on a 3-point or 5-point Likert scale ranging from. It consists of physical and emotional scales. Scores for each scale are calculated by using an algorithm and scores are standardized using a T-score metric with a mean of 50 and standard deviation of 10. Higher scores indicate better health-related quality of life.
Time Frame: 9 weeks after baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 11 | 13 | 14
T-score | .70 (5.66) | 1.91 (6.77) | -3.18 (10.12) | .50 (7.23)

6. Secondary Outcome: Change in Perceived Stress
Description: Changes in perceived stress will be measured by the Perceived Stress Scale (PSS-4). The 4-item measure asses stress experienced in the last month on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Scores range from 0-16, with higher scores indicating more stress.
Time Frame: 9 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 11 | 13 | 14
score on a scale | 1.23 (2.49) | .27 (2.41) | .15 (2.54) | 1.86 (2.44)

7. Secondary Outcome: Change in Stroke Knowledge
Description: Change in stroke knowledge will be measured by the Stroke Knowledge Instrument developed by the National Institutes of Health. This 7-item tool consists of true/false and multiple choice responses. Scores range from 0-7, with higher scores indicating more stroke knowledge.
Time Frame: 9 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 11 | 13 | 14
score on a scale | -.15 (1.34) | .27 (1.01) | .15 (1.34) | .29 (.99)

8. Secondary Outcome: Changes in Problem-Solving Abilities
Description: Changes in problem-solving abilities will be measured by the Social Problem-Solving Inventory - Short Form (SPSI-SF). The SPSI-SF is a 25-item tool consisting of five subscales (problem-solving orientation, rational problem-solving, negative problem-solving, impulsivity, avoidance style problem solving). Raw scores must first be converted to standard scores, which range from 0-20 for each of the 5 subscales. Higher scores on the problem-solving orientation and rational problem-solving scales indicate better problem-solving abilities, while higher scores on the negative problem-solving, impulsivity, and avoidance-style problem solving indicate worse problem-solving abilities. Total scores range from 0-100 with higher scores indicating better problem-solving abilities.
Time Frame: 9 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 11 | 13 | 14
score on a scale | 4.31 (12.28) | 4.55 (8.24) | 3.92 (6.98) | -1.07 (9.45)

9. Secondary Outcome: Caregiving Self-efficacy
Description: Changes in caregiving self-efficacy will be measured by the Caregiver Self-Efficacy Scale. This 14-item tool measures caregivers' judgments regarding their ability to perform effectively. Responses are binary (0=no, 1=yes) and scores range from 0-14, with higher scores indicating greater self-efficacy.
Time Frame: 9 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 11 | 13 | 14
score on a scale | -.23 (1.54) | .18 (3.54) | .77 (2.17) | -.71 (1.07)

10. Secondary Outcome: Change in Veteran Functional Abilities
Description: Change in Veteran functional abilities will be measured by the Barthel Index, which measures patients' abilities to perform 10 self-care tasks. Response options vary for each item and are scored on 5-point increments (e.g., 0=unable, 5=needs help, 10-independent). Total scores range from 0-100 with higher scores indicating greater functional abilities.
Time Frame: 9 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 11 | 13 | 14
score on a scale | -1.92 (14.51) | 2.27 (9.32) | 4.62 (9.23) | 1.43 (11.17)

11. Secondary Outcome: Change in Health-Related Quality of Life - Physical Scale
Description: Changes in health-related quality of life will be measured by the Rand 12-item Health Survey (VR-12). The VR12 items are scored on a 3-point or 5-point Likert scale ranging from. It consists of physical and emotional scales. Scores for each scale are calculated by using an algorithm and scores are standardized using a T-score metric with a mean of 50 and standard deviation of 10. Higher scores indicate better health-related quality of life.
Time Frame: 25 weeks after baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 10 | 13 | 13
T-score | -.48 (8.14) | 1.11 (8.96) | -7.50 (13.19) | .16 (5.87)

12. Secondary Outcome: Change in Perceived Stress
Description: Changes in stress will be measured by the Perceived Stress Scale (PSS-4). The 4-item measure asses stress experienced in the last month on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Scores range from 0-16, with higher scores indicating more stress.
Time Frame: 25 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 10 | 13 | 13
score on a scale | .92 (2.60) | .10 (2.42) | .54 (2.99) | 1.15 (2.12)

13. Secondary Outcome: Change in Stroke Knowledge
Description: as for outcome 7
Time Frame: 25 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 10 | 13 | 13
score on a scale | -.08 (1.50) | -.20 (.79) | -.08 (1.50) | .15 (.69)

14. Secondary Outcome: Change in Problem-Solving Abilities
Description: as for outcome 8
Time Frame: 25 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 10 | 13 | 13
score on a scale | 3.15 (11.26) | 7.40 (10.84) | -1.77 (8.57) | -1.08 (10.67)

15. Secondary Outcome: Change in Caregiving Self-Efficacy
Description: Changes in caregiving self-efficacy are measured by the Caregiver Self-Efficacy Scale. This 14-item tool measures caregivers' judgments regarding their ability to perform effectively. Responses are binary (0=no, 1=yes) and scores range from 0-14, with higher scores indicating greater self-efficacy.
Time Frame: 25 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 10 | 13 | 13
score on a scale | -.23 (1.83) | .20 (.92) | .38 (2.57) | -.62 (1.94)

16. Secondary Outcome: Change in Veteran Functional Abilities
Description: as for outcome 10
Time Frame: 25 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 10 | 13 | 13
score on a scale | -3.85 (21.42) | 4.00 (12.20) | 2.31 (14.52) | 0.00 (16.96)

17. Secondary Outcome: Change in Health-Related Quality of Life - Mental Scale
Description: as for outcome 11
Time Frame: 9 weeks after baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 11 | 13 | 14
T-score | -1.28 (9.86) | .09 (7.11) | 2.30 (10.41) | -1.98 (8.35)

18. Secondary Outcome: Change in Health-Related Quality of Life - Mental Scale
Description: as for outcome 11
Time Frame: 25 weeks after baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
Number analyzed (Participants) | 13 | 10 | 13 | 13
T-score | 1.44 (7.74) | -1.47 (10.62) | -4.32 (16.77) | -.99 (8.37)

ADVERSE EVENTS:
Arm/Group | 4-Week Intervention | 8-Week Intervention | 8-Week Attention Control | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/13 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4-Week Intervention (N=13) | 8-Week Intervention (N=13) | 8-Week Attention Control (N=13) | Standard Care (N=14)
Seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Caregiver reported they had a 2-day hospital stay for seizures related to dialysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes